CLINICAL TRIAL: NCT07167706
Title: Sleep Difficulties After Loss (SLEEPLOSS): Exploring the Beneficial Effect of Brief Behavioral Therapy for Insomnia in a Sample of Bereaved Individuals
Brief Title: Sleep Difficulties After Loss: Exploring the Beneficial Effect of Brief Behavioral Therapy for Insomnia in a Sample of Bereaved Individuals
Acronym: SLEEPLOSS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 116242
Record Dates: First submitted 2025-09-04; First posted 2025-09-11 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-08

CONDITIONS: Insomnia; Insomnia Chronic; Complicated Grief
Keywords: Insomnia; Insomnia Chronic; Brief Behavioral Therapy for Insomnia; BBTI; Sleep; Sleep Quality; Complicated Grief; Grief; Bereavement; Complicated Grief Reactions
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial with two arms. Participants are randomized to either an intervention group receiving BBTI or an an intervention group receiving sleep hygiene. The sleep hygiene group functions as an active control group, as sleep hygiene is not expected to improve sleep.
Who Masked: Participant
Masking Description: We aim to mask the participants as much as possible. The study uses a single-blind randomized controlled design, in which participants will know what treatment they will receive and that there are two groups. However, they will not know what treatment the other group will receive or that one group is the intervention group and the other an active control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (group 1) (Experimental): Participants will retrieve individually administered BBTI by therapists through face-to-face meetings and phone-calls. Treatment will take 4 weeks.
  Interventions: Behavioral: Brief Behavioral Therapy for Insomnia
- Active control group (group 2) (Sham Comparator): Participants will receive access to sleep hygiene education (SHE) through written educational material. Treatment will take 4 weeks.
  Interventions: Behavioral: Sleep Hygiene Therapy

INTERVENTIONS:
Behavioral: Brief Behavioral Therapy for Insomnia — BBTI is a multi-component intervention consisting of techniques from sleep restriction and stimulus control therapy. It targets behavioral elements of insomnia using four techniques: 1) reduce time in bed, 2) get up at the same time every day, 3) do not go to bed unless sleepy, and 4) do not stay in bed unless asleep.
  Other Names: BBTI
  Arms: Intervention group (group 1)
Behavioral: Sleep Hygiene Therapy — SHE consists of education on lifestyle factors (diet, exercise, substance use) and enviromental variables (noise, light, temperature) affecting sleep quality.
  Arms: Active control group (group 2)

SUMMARY:
The goal of the study is to investigate whether a brief behavioral therapy for insomnia (BBTI) improves sleep in bereaved patients screened for insomnia compared to an active control group (sleep hygiene education). The study will also explore if BBTI improves symptoms of complicated grief. The investigators will recruit approximately 58 bereaved participants with insomnia.

DETAILED DESCRIPTION:
The study is a randomized controlled trial comparing the effect of a brief behavioral therapy for insomnia (BBTI) on insomnia with an active control group (sleep hygiene). Participants will be 58 bereaved individuals who experience insomnia. After baseline assessment, participants will be randomized to either BBTI or sleep hygiene (active control). Both groups will undergo post-treatment assessments as well as 3- and 6-months follow-up assessments. The primary outcomes will be insomnia assessed with the Insomnia Severity Index (ISI) and improvements in sleep quality using the Pittsburgh Sleep Quality Index (PSQI) and sleep parameters using the consensus sleep diary. The secondary outcome will be complicated grief reactions (CGR) using the Aarhus Prolonged Grief Disorder scale (A-PGDs, prolonged grief). the Center of Epidemiological Studies Depression Scale (CESD-10, depression), the General Anxiety Disorder-7 questionnaire (GAD-7; anxiety), and the short-form PTSD Checklist for DSM-5 (PCL-5; PTSD).

The study has the following aims and hypotheses:

PRIMARY AIM: To investigate whether BBTI improves sleep in bereaved patients screened for insomnia when compared to an active control group.

PRIMARY HYPOTHESIS: Compared with the active control group, participants receiving BBTI will show statistically significant reductions in insomnia using the ISI, as well as improvements in sleep quality using the PSQI and sleep parameters using the consensus sleep diary.

SECONDARY AIM: To explore whether BBTI improves CGR in bereaved patients screened for insomnia when compared to an active control group.

SECONDARY HYPOTHESIS: Compared with the active control group, participants receiving BBTI will show statistically significant reductions in CGR using the A-PGDs, the CESD-10, the GAD-7, and the PCL-5.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Bereaved (experienced the death of a perceived loved one) ≥6 months ago
* Insomnia: a score of >10 on the Insomnia Severity index (ISI) and/or meet the Diagnostic and Statistical Manual of Mental Disorders, 5th Edition (DSM-5) criteria for Insomnia Disorder

Exclusion Criteria:

* Other sleep disor-ders (sleep apnea, parasomnia, narcolepsy)
* Use of drugs impacting sleep
* Severe psychological or physical disorders that may confound sleep (symptoms of CGR allowed)
* Neurodegenerative disorders
* Shift work
* Insufficient Danish proficiency
* Previous experience with BBTI or cognitive behavioral therapy for insomnia (CBT-I)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2025-12-30 (Estimated); Primary Completion 2027-05-31 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
Insomnia Severity Index (ISI) | Time Frame: Baseline (week 0), post-treatment (approximately week 4), 3-months follow-up (approximately week 16) 6-months follow-up (approximately week 28).
  The ISI measures the severity of insomnia symptoms and the associated impact on daytime functioning and distress. The questionnaire consists of 7 questions the sum of which makes up a total score. The ISI has a range of 0-28, with higher scores indicate worse insomnia severity.

SECONDARY OUTCOMES:
Pittsburgh Sleep Quality Index (PSQI) | Time Frame: Time Frame: Baseline (week 0), post-treatment (approximately week 4), 3-months follow-up (approximately week 16) 6-months follow-up (approximately week 28).
  Changes in sleep quality will be assessed using the Pittsburgh Sleep Quality Index (PSQI), with scores ranging from a minimum of 0, indicating no difficulty, to a maximum of 21, indicating severe difficulties in all areas related to sleep.
Consensus Sleep Diary | Time Frame: Time Frame: Baseline (week 0), post-treatment (approximately week 4), 3-months follow-up (approximately week 16) 6-months follow-up (approximately week 28).
  The Consensus Sleep Diary measures self-reported sleep providing various sleep parameters such as sleep duration, sleep onset latency (SOL), time in bed (TIB), total sleep time (TST), wake after sleep onset (WASO) and sleep efficiency (SE).
Morningness-Eveningness Questionnaire - Revised (MEQr) | Time Frame: Time Frame: Baseline (week 0)
  The Morningness-Eveningness Questionnaire-reduced (MEQr) will be used to assess circadian rhythm preferences (chronotype). This 5-item questionnaire evaluates sleep-wake patterns, preferred activity times, and subjective alertness at different times of the day. Scores categorize individuals as morning types, evening types, or intermediate types, with higher scores indicating a preference for morningness and lower scores indicating a preference for eveningness.
Aarhus Prolonged Grief Disorder Scale (A-PGDs) | Time Frame: Time Frame: Baseline (week 0), post-treatment (approximately week 4), 3-months follow-up (approximately week 16) 6-months follow-up (approximately week 28).
  The A-PGDs is a validated self-report instrument that will be used to measure symptoms of prolonged grief disorder, including yearning, emotional pain, difficulty moving on, and functional impairment. Items are rated on a Likert scale, and higher scores reflect more severe grief symptoms.
Center for Epidemiological Studies Depression Scale - 10 Item Version (CESD-10) | Baseline (week 0), post-treatment (approximately week 4), 3-months follow-up (approximately week 16), 6-months follow-up (approximately week 28).
  The CESD-10 is a short self-report questionnaire that will be used to measure the frequency of depressive symptoms over the past week. Scores range from 0 to 30, with higher scores indicating greater depressive symptom severity.
Generalized Anxiety Disorder - 7 Item Scale (GAD-7) | Baseline (week 0), post-treatment (approximately week 4), 3-months follow-up (approximately week 16), 6-months follow-up (approximately week 28).
  The GAD-7 will be used to measure generalized anxiety symptoms. It consists of 7 items rated on a 4-point Likert scale. Total scores range from 0 to 21, with higher scores reflecting greater anxiety severity.
PTSD Checklist for DSM-5 - Short Form (PCL-5 - Short Form) | Baseline (week 0), post-treatment (approximately week 4), 3-months follow-up (approximately week 16), 6-months follow-up (approximately week 28).
  The PCL-5 - Short Form is an abbreviated version of the PTSD Checklist that assesses core symptoms of post-traumatic stress disorder based on DSM-5 criteria. Items are rated on a Likert scale, with higher scores indicating greater PTSD symptom severity.
My Grief | Baseline (week 0), post-treatment (approximately week 4), 3-months follow-up (approximately week 16), 6-months follow-up (approximately week 28).
  MyGrief is a self-report questionnaire designed to evaluate grief-related symptoms and coping, specifically in relation to bereavement. It includes 33 items on emotional, cognitive, and functional aspects of grief, with higher scores reflecting greater grief-related difficulties.
The perceived stress scale (PSS) | Baseline (week 0), post-treatment (approximately week 4), 3-months follow-up (approximately week 16), 6-months follow-up (approximately week 28).
  The Perceived Stress Scale (PSS) will be used to measure the perception of stress. This 10-item questionnaire assesses how unpredictable, uncontrollable, and overloaded respondents find their lives. Higher scores indicate higher levels of perceived stress.
The Short-Form (12) Health Survey (SF-12) | Time Frame: Baseline (week 0), post-treatment (approximately week 4), 3-months follow-up (approximately week 16), 6-months follow-up (approximately week 28).
  The Short-Form (12) Health Survey (SF-12) will be used to assess health-related quality of life. This questionnaire comprises 12 items that evaluate eight domains of health: physical functioning, role limitations due to physical health problems, bodily pain, general health perceptions, vitality (energy/fatigue), social functioning, role limitations due to emotional problems, and mental health (psychological distress and well-being). Scores from these domains are combined to yield two summary measures: the Physical Component Summary (PCS) and the Mental Component Summary (MCS). Higher scores indicate better health-related quality of life across the evaluated domains.
World Health Organization-Five Well-Being Index (WHO-5) | Baseline (week 0), post-treatment (approximately week 4), 3-months follow-up (approximately week 16), 6-months follow-up (approximately week 28).
  The WHO-5 is a brief measure of subjective psychological well-being, consisting of 5 positively worded items. Higher scores indicate better well-being.
NEO Personality Inventory - Revised (NEO-PI-R), Neuroticism Only | Baseline (week 0)
  The Neuroticism domain of the NEO-PI-R assesses the tendency to experience negative emotions such as anxiety, anger, and depression. It is a self-report measure derived from the full NEO-PI-R personality inventory. Higher scores indicate greater neuroticism.
Experiences in Close Relationships Scale - Short Form (ECR-S) | Baseline (week 0)
  The ECR-S is a 12-item self-report questionnaire that measures adult attachment patterns, specifically attachment anxiety and attachment avoidance in close relationships. Higher scores reflect higher levels of attachment insecurity.
Expectancy/Credibility Questionnaire (CEQ) | Baseline (week 0)
  Treatment expectancy and rationale credibility will be measured with the Expectancy/Credibility Questionnaire (CEQ). Scores for each question range from 1 to 9 or 0% to 100%, with higher scores indicating greater treatment expectancy and credibility.

CONTACTS AND LOCATIONS:
Overall Officials: Alexander D Castro-Pavlik, PhD-student, MSc in Psychology, Principal Investigator — University of Aarhus
Locations (1):
- Aarhus University, Aarhus, Jutland, Denmark

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (e.g., outcome measure data underlying published analyses) will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 6 months after publication of the primary results and continuing for 5 years thereafter.
Access Criteria: Data will be made available to qualified researchers upon reasonable request to the study investigators, subject to approval and in accordance with applicable ethical and legal requirements.